CLINICAL TRIAL: NCT05878145
Title: Study on the Safety and Effectiveness of a Rehabilitation Exercise Program for Community-based Spinal Cord Injury Patients
Brief Title: Study on Rehabilitation Exercise Program for Community-based Spinal Cord Injury Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Sungchul Huh, Assistant professor, Pusan National University Yangsan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SCI REHAB EXERCISE RCT
Record Dates: First submitted 2023-04-27; First posted 2023-05-26 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Spinal Cord Injuries; Rehabilitation; Exercise Program
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): A 20-session structured rehabilitation exercise program in those with spinal cord injuries
  Interventions: Behavioral: Structured rehabilitation exercise program
- Control group (No Intervention): No exercise intervention in those with spinal cord injuries

INTERVENTIONS:
Behavioral: Structured rehabilitation exercise program — Stretching (10 mins): neck, shoulder, wrist, back; Aerobic exercise (20 mins): cycle ergometer, wheelchair run; Strengthening exercise (15 mins): shoulder press, chest press, front raise, biceps curl, lateral raise, bent over rowing or rowing, bent over lateral raise, triceps extension; Balance training (5 mins); Stretching exercise (10 mins)
  Arms: Intervention group

SUMMARY:
In the case of spinal cord injury, patients have shown a passive attitude towards participating in leisure sports or exercise programs, and there is a lack of suitable guidelines or experience in the local community for coaching exercise and sports for spinal cord injury patients, which makes coaches feel burdened when coaching these patients. Therefore, in this study, a suitable comprehensive exercise program will be designed and prescribed for patients who reside in the local community and want to participate in leisure sports, and the effectiveness and safety of the program will be verified. Based on the results, the aim of the study is to provide evidence that spinal cord injury patients can exercise safely and confidently in the local community in the future.

DETAILED DESCRIPTION:
Spinal cord injury is classified into complete paralysis and incomplete paralysis depending on the degree of spinal cord damage. In the case of complete paralysis, functional recovery is almost impossible, but in the case of incomplete paralysis, the level of functional recovery is determined through active rehabilitation exercises. In the past, most spinal cord injuries were traumatic, but due to the decrease in accidents, traumatic spinal cord injuries have decreased, and the incidence of non-traumatic spinal cord injuries (spinal cord disorders) has increased significantly due to aging. Most people with spinal cord injuries have difficulty performing appropriate rehabilitation exercises in the local community due to mobility impairments and limitations in daily activities. Spinal cord injury patients who participate in existing disabled sports are limited to some (relatively young) patients who have received epilepsy diagnosis. Individualized rehabilitation exercises based on each patient's personalized protocol are necessary, and sufficient functional recovery can be achieved through this approach. It is predicted that rehabilitation exercises through a protocol will improve cardiac and respiratory function and quality of life. Rehabilitation exercises for spinal cord injury patients should be applied based on accurate evaluation of function, and assessment of exercise-related risk factors should also be conducted. Customized exercise programs based on individual exercise function evaluations should be applied, but currently there is a lack of rehabilitation exercise programs that consider this. Additionally, risk factor evaluations related to exercise are not being conducted. Therefore, the development and application of patient-tailored community-based rehabilitation exercise programs for spinal cord injury patients that include risk factor evaluations and functional assessments are necessary.

ELIGIBILITY:
Inclusion Criteria:

* Spinal cord injury patients who are 19 years old or above and residing in the local community
* A person who can walk independently for more than 10 meters without assistance from others

Exclusion Criteria:

* Individuals who have difficulty understanding the exercise program or expressing their symptoms
* Individuals who cannot participate in the intervention exercise program due to serious cardiovascular diseases
* Individuals who are deemed unsuitable for this study by a specialist in rehabilitation medicine due to other medical conditions

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2023-05-27 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
EuroQol 5 Dimension 5 Level | Baseline evaluation and follow-up evaluation immediately after average 2 months of exercise program
  Self-report survey that measures quality of life across 5 domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Converting the patient's response results using quality weights has a value between 0.000 and 1.000. A higher score means a higher quality of life.
6 minute walk distance | Baseline evaluation and follow-up evaluation immediately after average 2 months of exercise program
  Sub-maximal exercise test used to assess aerobic capacity and endurance. Longer distances indicate better athletic ability.

SECONDARY OUTCOMES:
Spinal cord independence measure III | Baseline evaluation and follow-up evaluation immediately after average 2 months of exercise program
  Tool to evaluate independence of spinal cord injury patients. The total score ranges from 0 to 100, and the higher the score, the more independent the patient is.
Berg balance scale | Baseline evaluation and follow-up evaluation after average 2 months of exercise program
  Testing tool with high validity and reliability used to measure balance. Each item is scored 0-4 points, with a total score of 0-56 points. A higher score means better balance ability.
Timed up and go test | Baseline evaluation and follow-up evaluation immediately after average 2 months of exercise program
  Reliable and valid test for quantifying functional mobility. The time it takes for a patient to get up from a chair, walk 3 meters, and come back to sit down is measured. The shorter the time, the better the mobility.
Grip strength | Baseline evaluation and follow-up evaluation immediately after average 2 months of exercise program
  Force applied by the hand to pull on or suspend from objects. It is widely used to assess sarcopenia and as a surrogate indicator of muscle strength. Measured in kg, the higher the value, the stronger the grip is considered.
30 second sit to stand test | Baseline evaluation and follow-up evaluation immediately after average 2 months of exercise program
  Testing leg strength and endurance. It measures the number of times a person can stand up from a chair and sit down again in 30 seconds, and the higher the number, the better function and strength.
Sit and reach test | Baseline evaluation and follow-up evaluation immediately after average 2 months of exercise program
  Test to measure hamstring and low back flexibility. It is expressed in centimeters (cm), and if the fingertips touch in front of the toes, it is recorded as a positive number (+), and if the fingertips touch behind the toes, it is recorded as a negative number (-).
Beck anxiety inventory | Baseline evaluation and follow-up evaluation immediately after average 2 months of exercise program
  Anxiety measuring tool. Each item is scored 0-3 points, with a total score of 0-63 points. A score of 0-7 indicates minimal anxiety, a score of 8-15 indicates mild anxiety, a score of 16-25 indicates moderate anxiety, and a score of 26-63 indicates severe anxiety.
Beck depression inventory | Baseline evaluation and follow-up evaluation immediately after average 2 months of exercise program
  Depression measuring tool. Each item is scored 0-3 points, with a total score of 0-63 points. A score of 0-13 indicates minimal depression, a score of 14-19 indicates mild depression, a score of 20-28 indicates moderate depression, and a score of 29-63 indicates severe depression.
Fat-free mass from bioelectrical impedance analysis | Baseline evaluation and follow-up evaluation immediately after average 2 months of exercise program
  A method used to measure the components of the body. It is the total amount (kg) of body components excluding body fat, and the higher it is, the better the body composition is interpreted.
Fat-free mass index from bioelectrical impedance analysis | Baseline evaluation and follow-up evaluation after average 2 months of exercise program
  A method used to measure components of the body. This is an indicator that standardizes fat-free mass according to body size. The higher it is, the more muscle mass and the better health.
Percent body fat from bioelectrical impedance analysis | Baseline evaluation and follow-up evaluation immediately after average 2 months of exercise program
  A method used to measure the components of the body. The normal range varies depending on age and gender. The lower the score within the general normal range, the better the health. The higher it is, the higher the risk of obesity-related diseases.
skeletal muscle mass from bioelectrical impedance analysis | Baseline evaluation and follow-up evaluation immediately after average 2 months of exercise program
  A method used to measure the components of the body. Normal range varies depending on age and gender. The higher it is within the general normal range, the better the health. The lower it is, the higher the risk of lack of strength and sarcopenia.

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Hwa Ko, PhD, Principal Investigator — Pusan National University Yangsan Hospital
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huh S, Kim Y, Ko HY, Yun MS, Shin YI, Lee JL, Ko SH. Effectiveness of a Community-Based Exercise Program for Ambulatory Individuals With Spinal Cord Injury: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2025 Apr;106(4):481-490. doi: 10.1016/j.apmr.2024.11.003. Epub 2024 Nov 21. PMID 39577713